CLINICAL TRIAL: NCT01679951
Title: A Phase 2b Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel Group, Dose Range Finding Study of JNJ-38518168 in Subjects With Active Rheumatoid Arthritis Despite Concomitant Methotrexate Therapy
Brief Title: A Dose Range Finding Study of JNJ-38518168 in Patients With Active Rheumatoid Arthritis in Spite of Treatment With Methotrexate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision was made to prematurely discontinue this trial due to lack of efficacy.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100734; 38518168ARA2002 (Other: Janssen Research & Development, LLC); 2011-002840-29 (EudraCT Number)
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Swollen and tender joints; Methotrexate; Immunology; Dose range finding study
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Methotrexate
- JNJ-38518168 (3 mg/d) (Experimental)
  Interventions: Drug: JNJ-38518168 (3 mg); Drug: Methotrexate
- JNJ-38518168 (10 mg/d) (Experimental)
  Interventions: Drug: JNJ-38518168 (10 mg); Drug: Methotrexate
- JNJ-38518168 (30 mg/d) (Experimental)
  Interventions: Drug: JNJ-38518168 (30 mg); Drug: Methotrexate

INTERVENTIONS:
Drug: Placebo — Form=tablet, route=oral. Placebo will be administered once daily from week 0 to week 24.
  Arms: Placebo
Drug: JNJ-38518168 (3 mg) — Type=exact number, unit=mg, number=3, form=tablet, route=oral. JNJ-38518168 will be administered once daily up to 24 weeks.
  Arms: JNJ-38518168 (3 mg/d)
Drug: JNJ-38518168 (10 mg) — Type=exact number, unit=mg, number=10, form=tablet, route=oral. JNJ-38518168 will be administered once daily up to 24 weeks.
  Arms: JNJ-38518168 (10 mg/d)
Drug: JNJ-38518168 (30 mg) — Type=exact number, unit=mg, number=30, form=tablet, route=oral. JNJ-38518168 will be administered once daily up to 24 weeks.
  Arms: JNJ-38518168 (30 mg/d)
Drug: Methotrexate — Participants must have been treated with and tolerated Methotrexate (MTX) treatment at dosages from 10 to 25 milligram per week (mg/week) inclusive, for a minimum of 6 months prior to the date of signing the informed consent at screening and must have a stable MTX dose for a minimum of 8 weeks prior to the date of signing the informed consent at screening and continue to receive the same MTX dose at Week 0 through Week 24.

SUMMARY:
The purpose of this dose range finding study is to assess the effectiveness, safety and tolerability of JNJ-38518168 at doses of 3, 10, and 30 mg/d compared with placebo in patients with active rheumatoid arthritis (RA) despite concomitant methotrexate (MTX) therapy.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor patient knows the treatment that the patient receives), multicenter, placebo-controlled (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), parallel-group (each group of patients will be treated at the same time), dose range finding study of JNJ-38518168 in patients with active RA despite concomitant MTX therapy. The study will consist a screening period, a 24-week placebo-controlled period and a 4-week follow-up period between the last dose and the last visit. The duration of participation in the study for an individual patient will be up to 34 weeks (including screening). The patients will be assigned to 1 of 4 treatment groups in a 1:1:1:1 ratio to placebo and JNJ-38518168 (3 mg or 10 mg or 30 mg). Safety assessments and evaluations to determine the efficacy of JNJ-38518168 to reduce the signs and symptoms of RA will be performed at study visits. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Has had rheumatoid arthritis for at least 6 months prior to the date of signing the informed consent at screening
* Must be positive for either anti-cyclic citrullinated peptide antibody or rheumatoid factor in serum at screening
* Must have active rheumatoid arthritis (at least 6 swollen and 6 tender joints using a 66/68 joint count at the time of screening and at baseline and Serum C reactive protein greater than or equal to 0.80 mg/dL at the time of screening
* Has been treated with and tolerated methotrexate treatment at dosages from 10 to 25 mg/week inclusive, for a minimum of 6 months with stable dose for at least 8 weeks prior to the date of signing the informed consent at screening

Exclusion Criteria:

* Has inflammatory diseases other than rheumatoid arthritis, including but not limited to adult onset Still's disease, psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, and Lyme disease that might confound the evaluation of the benefit of study agent therapy
* Has current signs or symptoms of liver or renal insufficiency or cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances that are severe, progressive or uncontrolled
* Has ever received any approved or investigational biologic agent for a rheumatoid indication
* Has been treated with any nonbiologic disease modifying antirheumatic drugs within 4 weeks prior to the first administration of study agent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2014-04-17 (Actual); Study Completion 2014-07-03 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score 28 (DAS28) (C-reactive protein [CRP]) at Week 12 | Baseline and Week 12
  The DAS28 using CRP is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP, and Patient's Global Assessment of Disease Activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst.

SECONDARY OUTCOMES:
Change from baseline in DAS28 (CRP) at Week 24 | Baseline and Week 24
Change from baseline in DAS28 (erythrocyte sedimentation rate [ESR]) at Week 12 and Week 24 | Baseline, Week 12 and Week 24
DAS28 (CRP) response rates at Week 12 and Week 24 | Week 12 and Week 24
DAS28 (ESR) response rates at Week 12 and Week 24 | Week 12 and Week 24
DAS28 (CRP) remission rates at Week 12 and Week 24 | Week 12 and Week 24
DAS28 (ESR) remission rates at Week 12 and Week 24 | Week 12 and Week 24
American College of Rheumatology (ACR) 20/50/70 response rates at Week 12 and Week 24 | Week 12 and Week 24
  An ACR 20/50/70 response is defined as a greater than or equal to 20/50/70 percentage improvement from baseline in: 1. Swollen joint count (66 joints) and tender joint count (68 joints) 2. greater than or equal to 50 percentage improvement in 3 of the following 5 assessments: a. Patient's assessment of pain (VAS) (0-10 cm) b.Patient's Global Assessment of Disease activity (VAS) (0-10 cm) c. Physician's Global Assessment of Disease Activity (VAS) (0-10 cm) d. Patient's assessment of physical function as measured by the Health Assessment Questionnaire (HAQ) e. C reactive protein (CRP).
Hybrid ACR response at Week 12 and Week 24 | Week 12 and Week 24
  The hybrid ACR response is a continuous variable that is limited to an overall score of -100 (maximal worsening) to +100 (maximal improvement).
ACR/European League Against Rheumatism (EULAR) remission rates at Week 12 and Week 24 | Week 12 and Week 24
  According to the ACR/EULAR provisional definition, a patients RA can be defined as being in remission based on either of 2 definitions:
  when scores on the tender joint count, swollen joint count, CRP (in mg/dL), and patient global assessment (0-10 scale) are all less than or equal to 1 OR when the score on the simplified disease activity index (SDAI) is less than or equal to 3.3 Analyses based on each definition will be performed.
Change from baseline in Simplified Disease Activity Index (SDAI) at Week 12 and Week 24 | Baseline, Week 12 and Week 24
  The SDAI is the numerical sum of 5 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, patient global assessment of disease activity (PGA VAS in cm), physician global assessment of disease activity (MDGA VAS in cm) and C-reactive protein (CRP in mg/dL).
Change from baseline in Clinical Disease Activity Index (CDAI) at Week 12 and Week 24 | Baseline, Week 12 and Week 24
  The CDAI is the numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA, and MDGA.
Health Assessment Questionnaire - Disability Index (HAQ-DI) response at Week 12 and Week 24 | Week 12 and Week 24
  The HAQ-DI is a 20-question instrument that assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty), to 3 (inability to perform a task in that area).
Change from baseline in HAQ-DI score at Week 12 and Week 24 | Baseline, Week 12 and Week 24
Percent change from baseline in ESR levels at Week 12 and Week 24 | Baseline, Week 12 and Week 24
Percent change from baseline in ACR components at Week 12 and Week 24 | Baseline, Week 12 and Week 24
Number of patients with adverse events | Up to Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (85):
- United States (9):
  - Huntsville, Alabama
  - Gilbert, Arizona
  - Covina, California
  - Palm Harbor, Florida
  - Granger, Indiana
  - Frederick, Maryland
  - Freehold, New Jersey
  - Charlotte, North Carolina
  - Charleston, South Carolina
- Argentina (2):
  - Buenos Aires
  - San Miguel de Tucumán
- Chile (4):
  - Osorno X Region
  - Santiago
  - Santiago - Macul
  - Viña del Mar
- Colombia (5):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Cali
  - Medellín
- Czechia (5):
  - Hlučín
  - Ostrava
  - Prague
  - Slaný
  - Zlín
- Hungary (5):
  - Balatonfüred
  - Budapest
  - Debrecen
  - Gyulai
  - Veszprém
- Japan (13):
  - Chiba
  - Fukuoka
  - Hokkaido
  - Kanagawa
  - Katō
  - Kawagoe
  - Kumamoto
  - Kyoto
  - Matsuyama
  - Osaka
  - Sapporo
  - Takasaki
  - Tokyo
- Latvia (3):
  - Ādaži
  - Riga
  - Valmiera
- Mexico (9):
  - Del Gustavo A Madero
  - Delegación Cuauhtémoc
  - Guadalajara
  - Guadalajara, Jalisco
  - Guadalaja
  - León
  - Mexico City
  - México
  - San Luis Potosí City
- Poland (7):
  - Bialystok
  - Katowice
  - Nadarzyn
  - Poznan
  - Środa Wielkopolska
  - Warsaw
  - Wroclaw
- Romania (4):
  - Bacau
  - Brăila
  - Bucharest
  - Sibiu
- Russia (8):
  - Kazan'
  - Moscow
  - Novosibirsk
  - Petrozavodsk
  - Saint Petersburg
  - Saratov
  - Tver'
  - Yaroslavl
- South Korea (3):
  - Daegu
  - Pucheon
  - Suwon
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- Thailand (2):
  - Bangkok
  - Chiang Mai
- Ukraine (3):
  - Donetsk
  - Kyiv
  - Vinnytsia